CLINICAL TRIAL: NCT03451630
Title: Leveraging Integrated Models of Care to Improve Patient-Centered Outcomes for Publicly-Insured Adults With Complex Health Care Needs
Brief Title: Integrated Care (IC) Models for Patient-Centered Outcomes
Acronym: IC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Daniel Swayze, Vice President, Community Services for UPMC Health Plan, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY19030130; IHS-1609-36670 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2018-01-30; First posted 2018-03-02 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Diabetes; Asthma; Chronic Obstructive Pulmonary Disease; Hypertension; Anxiety; Atrial Fibrillation; Congestive Heart Failure; Depression; Bipolar Disorder; Schizophrenia
Keywords: chronic conditions; care management; digital tools
MeSH Terms: conditions — Diabetes Mellitus; Asthma; Pulmonary Disease, Chronic Obstructive; Hypertension; Anxiety Disorders; Atrial Fibrillation; Heart Failure; Depression; Bipolar Disorder; Schizophrenia; Chronic Disease

STUDY DESIGN:
Intervention Model Description: We chose an individual, stratified randomized trial design to randomly assign each enrollee to one of the three interventions arms, minimizing and balancing confounding variables. We will utilize an unequal randomization ratio of 2:2:1 for High-Touch, High-Tech, and ODP, respectively. While the less resource intensive ODP, in fact, improve meaningful outcomes for certain patient subgroups, our health care system has invested heavily in High-Touch and High-Tech as evidence-based solutions for chronic disease care. We will use a mixed-methods approach that incorporates both qualitative and quantitative data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Touch (Active Comparator): Delivered primarily via face-to-face interactions, with telephonic interactions and information sharing that does not require access to mobile devices or the Internet. In-person support and/or telephonic interactions to occur at least four times over at least a four-month period.
  Interventions: Behavioral: High-Touch
- High-Tech (Active Comparator): Delivered via a remote care management platform and digital health tools. Remote care support interactions to occur for at least a four-month period.
  Interventions: Behavioral: High-Tech
- Optimal Discharge Planning (Active Comparator): Delivered via Health Plan support and resources within 14-30 days of an initial home or telephonic visit.
  Interventions: Behavioral: Optimal Discharge Planning

INTERVENTIONS:
Behavioral: High-Touch — Intensive, in-person and/or telephonic support.
  Arms: High-Touch
Behavioral: High-Tech — Remote care management and self-directed digital tools.
  Arms: High-Tech
Behavioral: Optimal Discharge Planning — Transition to other Health Plan disease management programs and/or community resources.
  Arms: Optimal Discharge Planning

SUMMARY:
Multiple chronic conditions (MCC) are widely recognized as the U.S. public health challenge of the 21st century. These physical and behavioral health conditions take a large toll on those living with chronic diseases, including many who are publicly insured, as well as caregivers and society. While evidence-based integrated care models can improve outcomes for individuals with MCC, such models have not yet been widely implemented. Insurance providers/payers have innovative system features that can be used to deploy these models; however, the investigators do not yet know which of these features can best help to improve outcomes for individuals with MCC in general or high-need subgroups in particular. As a result, patients lack information to make important decisions about their health and health care, and system-level decision makers face ongoing challenges in effectively and efficiently supporting those with MCC.

This real-world study will provide useful information about available options for supporting individuals with MCC. Building on existing integrated care efforts, the investigators will enroll N=1,400 (a modified total N) adults with MCC at risk for repeated hospitalizations and assess the impact of three payer-led options (e.g. High-Touch, High-Tech, Standard Care/Optimal Discharge Planning (ODP)) on patient-centered outcomes, namely patient activation in health care, health status, and subsequent re-hospitalization. The investigators will also determine which option works best for whom under what circumstances by gathering information directly from individuals with MCC through self-report questionnaires, health care use data, and interviews.

DETAILED DESCRIPTION:
Study aims. Given the documented need for valuable information about system-level features that can be used to effectively and efficiently support adults in living well with MCC, this study is designed to achieve the following aims:

Aim 1: Compare the effectiveness of High-Touch, High-Tech, and ODP on primary outcomes including hospital readmission, health status, and patient activation, and on several secondary outcomes including functional status, quality of life, care satisfaction, emergent care use, engagement in primary, specialty, and mental health care, and gaps in care.

Aim 2: Examine the differential effects of the interventions for patient subgroups, based on age, race, illness complexity, and comorbid behavioral health conditions to evaluate heterogeneity of treatment effects (HTE) and determine for whom and in what circumstances the interventions are most effective.

Aim 3: Examine perceived barriers and facilitators to efficient and effective implementation of High-Touch and High-Tech interventions for delivering evidence-based integrated care.

An individual-level randomized design along with a pragmatic, mixed-methods approach to compare system-level features for delivering evidence-based components of integrated care for Medicaid or dual-eligible adult members with MCC who reside in in Western, Central, or Eastern PA and are at high risk for rehospitalization has been selected for this study. This design, based on significant input from patient stakeholders and Drs. Kevin Kraemer (Scientific Co-I; health services researcher) and Doug Landsittel (Co-I; biostatistician/CER expert), accords fully with the PCORI Methodology Standards. Intervention effectiveness will be determined by examining the differential impact on outcomes that are most meaningful to patients in our target population and those delivering their care. The scope and duration of the study interventions and evaluation are sufficient to measure change in patient-centered outcomes.

High-Touch, High-Tech, and ODP will serve as the comparators for this study. ODP follows standardized procedures for patient engagement including when a patient is either hospitalized or transitioning from the hospital setting into ambulatory care for follow-up and condition management. Due to resources and other limitations, not all patients who are eligible for High-Touch/High-Tech enroll in these programs. Thus, the addition of the ODP arm will allow for a less intensive model to be examined and targeted to appropriate patient populations.

For Aims 1 and 2, an individual, stratified randomized trial design was selected to randomly assign each enrollee to one of the three interventions arms, minimizing and balancing for confounding variables. Individual-level randomization was selected as opposed to cluster randomization at a system level (e.g. practice-, hospital-level) because the interventions are delivered by a single payer and are not subject to within-practice contamination. Based on valuable system-level stakeholder feedback, an unequal randomization ratio of 2:2:1 for High-Touch, High-Tech, and ODP, respectively, was utilized. While the less resource intensive ODP may, in fact, improve meaningful outcomes for certain patient subgroups, the health care system has invested heavily in High-Touch and High-Tech as evidence-based solutions for chronic disease care. Additionally, stakeholders have indicated that they would like as many participants as possible to have a fully integrated care experience offered by High-Touch/High-Tech and would like to limit enrollment into ODP. The investigators will use a mixed-methods approach that incorporates both qualitative and quantitative data. The addition of qualitative data collection and analyses in Aim 3 will permit more comprehensive understanding of patient and staff experiences with the interventions and results will aide in dissemination of study findings in a manner that is most consistent with patient and other stakeholder perceptions and experiences. The overall, four-year study timeline includes three phases: Pre-Intervention (months 1-6), Intervention and Data Collection (months 7-40), and Data Analysis and Reporting (months 41-48). Note: a 19-month no cost extension was granted to the study team to complete enrollment and data collection, especially during workflow adaptations related to COVID-19 restrictions.

The study population includes Medicaid or dual-eligible (Medicare-Medicaid) adults age 21 years and older with MCC, including at least one physical health condition (e.g., cardiovascular disease, hypertension, COPD, diabetes) and at least one additional physical or behavioral health condition (e.g., depression, serious mental illness, substance abuse disorder) and at least one hospital discharge in the previous 30 days. These individuals will reside in PA and will be insured through physical and/or behavioral health payers within the UPMC Insurance Services Division (ISD). In addition, these individuals will have several comorbidities, will have been prescribed several medications, and/or will be predicted future high health care utilizers. Based on a 75% enrollment rate, we initially expected1,662 individuals to be randomized to either High-Tech (n=667), High-Touch (n=667) or ODP (n=328). However, our funder approved a sample size recalculation for an 90% retention rate for 1,400 consented individuals randomized to either High-Tech (n=448), High-Touch (n=448) or ODP (n=224).

The study will use web-based randomization to one of the three interventions for those individuals who consent to participate in the study. Once a member of the Community Team (CT), multidisciplinary community-based team of nurses, licensed social workers, and licensed professional counselors, determines eligibility, CT personnel will enter key identification information, and the system will then generate a Study ID (numeric identification number) along with assignment to an intervention arm. Randomization will be stratified by gender, type of insurance (Medicaid or Medicare-Medicaid), and technology/digital literacy, which will be assessed at time of enrollment and before randomization, to ensure that intervention arms are balanced with respect to these important variables. Within each stratum, random block sizes of 5 and 10 will be used to maximize balance between intervention groups while minimizing the ability to unmask investigators to the next treatment assignment, triggering an automated alert to CT staff regarding which intervention to implement for each participant and documented accordingly in HealthPlaNET, UPMC ISD's integrated health management software program. If a participant is unwilling to be randomized, they will be excluded from the study.

Each patient is assigned a care manager (CM) who provides comprehensive services for the duration of intervention implementation. Bilingual staff will be available to support native Spanish speaking participants. CMs are currently employed to develop and implement care plans with patients, coordinate healthcare services, work with the pharmacist to manage patient's medications, make home visits, and deliver telehealth care and remote monitoring.

Patients in both High-Touch and High-Tech will experience similar procedures at the start of their participation. A CM engages patients in a face-to-face assessment in-home or telephonically to dialogue about the social determinants affecting continued hospital readmissions and emergency department use. At the completion of the assessment, the study is presented to the member and if agreeable informed consent occurs. Individuals randomized to ODP will be provided with the transitional care services. High-Touch and High-Tech interventions are provided for four to twelve months following hospitalization, based on need, and ODP participants are transitioned to appropriate Health Plan or community resources within 14 to 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Medicaid or dual-eligible (Medicare-Medicaid) adults, ages 21 years and older with Multiple Chronic Conditions (MCC).
2. Have at least one physical health condition (e.g., cardiovascular disease, hypertension, COPD, diabetes).
3. Have at least one additional physical or behavioral health condition (e.g., depression, serious mental illness, substance abuse disorder).
4. Reside in Western, Central, or Eastern Pennsylvania.
5. Be insured through physical and/or behavioral health payers within the UPMC ISD.
6. Individuals will have several comorbidities, will have been prescribed several medications, and/or will be predicted future high health care utilizers.
7. Must have at least one hospital discharge within 30 days of enrollment.
8. Speak and read English or Spanish at a 4th grade level.

Exclusion Criteria:

1. Individuals receiving advanced levels of care, including:

   * Individuals who are pregnant.
   * Individuals in skilled nursing facilities or receiving hospice or palliative care.
   * Individuals on hemodialysis for kidney disease.
   * Individuals whose inpatient admission was related to active cancer treatment.
2. Individuals currently enrolled in an RPM program.
3. Individuals who have participated in High-Touch or High-Tech within the previous 12 months.
4. Individuals who are unable to operate a smart phone due to limitations in literacy, vision, or dexterity.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Swayze, DrPH, MBA, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the questions asked in this study, survey respondents were assured raw data would remain confidential and would not be shared.

REFERENCES:
- [Background] Kearney SM, Williams K, Nikolajski C, Park MJ, Kraemer KL, Landsittel D, Kang C, Malito A, Schuster J. Stakeholder impact on the implementation of integrated care: Opportunities to consider for patient-centered outcomes research. Contemp Clin Trials. 2021 Feb;101:106256. doi: 10.1016/j.cct.2020.106256. Epub 2020 Dec 29. PMID 33383229
- [Background] Williams K, Markwardt S, Kearney SM, Karp JF, Kraemer KL, Park MJ, Freund P, Watson A, Schuster J, Beckjord E. Addressing Implementation Challenges to Digital Care Delivery for Adults With Multiple Chronic Conditions: Stakeholder Feedback in a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Feb 1;9(2):e23498. doi: 10.2196/23498. PMID 33522981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between September 4, 2018 and November 4, 2021. Care Managers enrolled eligible individuals during an initial in-home or telephonic visit; a study team member conducted randomization.
Period: Overall Study
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Started | 562 | 552 | 286
Completed | 535 | 529 | 268
Not Completed | 27 | 23 | 18
Not completed — Death | 15 | 16 | 11
Not completed — Lost to Follow-up | 9 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Unable to confirm accurate eligibility criteria after randomization and intervention completion. | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Three participants formally withdrew from the High-Tech arm and are therefore excluded from the analysis. Additionally, we could not confirm accurate eligibility criteria for 10 participants at the time of analysis, so they are also excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning | Total
Number analyzed (Participants) | 559 | 545 | 283 | 1387
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.87 (11.68) | 53.59 (11.59) | 53.67 (12.08) | 53.32 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341 | 345 | 188 | 874
  Male | 218 | 200 | 95 | 513
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 9 | 39
  Not Hispanic or Latino | 544 | 530 | 274 | 1348
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 5 | 3 | 15
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 0 | 4
  Black or African American | 122 | 120 | 57 | 299
  White | 414 | 394 | 204 | 1012
  More than one race | 10 | 8 | 9 | 27
  Unknown or Not Reported | 4 | 15 | 10 | 29
Charlson Comorbidity Index (CCI) [Mean (Standard Deviation); unit: units on a scale] — The Charlson Comorbidity Index (age-adjusted) is designed to predict survival rates for patients with multiple comorbidities after a hospitalization. A scores range from 0 to 37, with a higher score indicating a higher mortality risk. We assess CCI based on the previous 12 months of claims.
  units on a scale | 4.94 (3.23) | 5.14 (3.07) | 5.16 (3.42) | 5.06 (3.21)
Area Deprivation Index (ADI) [Mean (Standard Deviation); unit: units on a scale] — The Area Deprivation Index (ADI) is a measure used to account for the impact of resources in a geographic area that influence an individual's health, such as income, education, employment, and housing quality. Available ADI data ranges from -48 to 129, with higher numbers indicating a more resourced area of residence.
  units on a scale | 109.64 (5.29) | 109.45 (5.62) | 109.60 (5.11) | 109.56 (5.38)
Comfort with Technology/ Digital Literacy [Count of Participants; unit: Participants]
  Comfortable: Disagree Strongly | 33 | 41 | 16 | 90
  Comfortable: Disagree | 85 | 70 | 35 | 190
  Comfortable: Agree | 310 | 296 | 162 | 768
  Comfortable: Agree Strongly | 131 | 138 | 70 | 339
Line of Business (Medicaid/ Medicaid-Medicare) [Count of Participants; unit: Participants]
  Medicare-Medicaid | 118 | 107 | 59 | 284
  Medicaid | 441 | 438 | 224 | 1103
Engagement at Baseline [Count of Participants; unit: Participants] — The definition of engagement is as follows:
  1. ODP Engagement: In-home or telephonic visit or video visit occurred within 1 week of initial visit
  2. High Touch Engagement: In-home or telephonic visit occurred within 4 weeks of the initial visit.
  3. High-Tech Engagement: Telephonic visit or video visit occurred within 4 weeks of Initial Visits.
  Note: Care activities also occurred outside of visits; a follow-up visit was not a requirement of ODP.
  Participants
    No | 215 | 213 | 246 | 674
    Yes | 344 | 332 | 37 | 713

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation
Description: Assessed using the Patient Activation Measure (PAM), a 13-item scale that gauges individual knowledge, skills, and confidence essential to managing one's own health. We assess a global score of the PAM measure, with scores ranging from 0 to 100; lower values represent a poor outcome while higher values represent a better outcome.
Time Frame: Baseline, 3-, 6-, and 12-months.
Population: Includes all individuals who completed the measure at least one timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 495 | 506 | 237
score on a scale
  Baseline | 61.87 (14.36) | 63.73 (16.10) | 63.82 (16.12)
  3-Months: number analyzed (Participants) | 457 | 480 | 228
  3-Months | 63.15 (15.56) | 63.60 (16.65) | 63.60 (15.98)
  6-Months: number analyzed (Participants) | 441 | 457 | 217
  6-Months | 62.55 (16.03) | 62.15 (15.84) | 64.76 (15.98)
  12-Months: number analyzed (Participants) | 441 | 448 | 218
  12-Months | 63.15 (15.05) | 64.58 (15.41) | 62.83 (15.75)
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall Test of Group by Time Interaction; Test type: Superiority; p = 0.0211, Mixed Models Analysis — Controlling for: age, sex, race, ethnicity, insurance, engagement at baseline, comfortability with technology, tech literacy (HINTS), social support at baseline (ISEL), health literacy (AAHLS), illness burden (CCI), and area deprivation index (ADI); F-statistics 2.49 with degrees of freedom (6, 3152)
Statistical Analysis 2: Comparison: High-Touch vs Optimal Discharge Planning; Test for group difference in the change from baseline to 12-Months using linear contrast; Test type: Superiority; p = 0.0280, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 4.83 with degrees of freedom (1, 3152); Mean Difference (Final Values) = 2.69, 95% CI 2-sided [0.29 to 5.09], Standard Error of Mean 1.22
Statistical Analysis 3: Comparison: High-Tech vs Optimal Discharge Planning; Test for group difference in the change from baseline to 12-Months using linear contrast; Test type: Superiority; p = 0.0935, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 2.81 with degrees of freedom (1, 3152); Mean Difference (Final Values) = 2.07, 95% CI 2-sided [-0.35 to 4.48], Standard Error of Mean 1.23
Statistical Analysis 4: Comparison: High-Touch vs High-Tech; Test for group difference in the change from baseline to12-Months using linear contrast; Test type: Superiority; p = 0.5538, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.35 with degrees of freedom (1, 3152); Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-1.44 to 2.68], Standard Error of Mean 1.05

2. Primary Outcome: Change in Health Status
Description: Assessed using the RAND 36-Item Short Form Survey 1.0 (SF-36). The SF-36 is a set of 36 health status and quality-of-life measures that are patient self-reported and measure functional health and well-being within eight domains, including physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. Values are recoded per the scoring key relating each item to the appropriate subscale. All items are scored so that a high score defines a more favorable health state. We assess a global scale with a 0 to 100 range with 0 being worst possible health status and 100 being the best possible health status.
Time Frame: Baseline, 3-, 6-, and 12-months.
Population: Includes all individuals who completed the measure at least one timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 496 | 505 | 236
score on a scale
  Baseline | 39.61 (18.39) | 39.50 (18.65) | 39.05 (17.80)
  3-Month: number analyzed (Participants) | 457 | 479 | 228
  3-Month | 42.12 (20.06) | 42.03 (19.90) | 41.31 (19.99)
  6-Month: number analyzed (Participants) | 440 | 455 | 215
  6-Month | 41.86 (19.84) | 41.39 (19.84) | 41.83 (20.84)
  12-Month: number analyzed (Participants) | 442 | 450 | 218
  12-Month | 42.68 (20.50) | 42.27 (19.63) | 40.85 (19.03)
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall Test of the Group by Time Interaction; Test type: Superiority — Controlling for: age, sex, race, ethnicity, insurance, engagement at baseline, comfortability with technology, tech literacy (HINTS), social support at baseline (ISEL), health literacy (AAHLS), illness burden (CCI), and area deprivation index (ADI); p = 0.8505, Mixed Models Analysis; F-statistics 0.44 with degrees of freedom (6, 3154)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for significant change over time when the treatment-by-time interaction effect is not significant; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 16.97 with degrees of freedom (3, 3160)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for significant change by treatment when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.8656, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.14 with degrees of freedom (2, 1229)
Statistical Analysis 4: Comparison: High-Touch vs Optimal Discharge Planning; Test for group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.4740, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.51 with degrees of freedom (1, 3154); Mean Difference (Final Values) = 0.93, 95% CI 2-sided [-1.61 to 3.46], Standard Error of Mean 1.29
Statistical Analysis 5: Comparison: High-Tech vs Optimal Discharge Planning; Test for group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.6017, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.27 with degrees of freedom (1, 3154); Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-1.81 to 3.13], Standard Error of Mean 1.26
Statistical Analysis 6: Comparison: High-Touch vs High-Tech; Test for group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.7860, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.07 with degrees of freedom (1, 3154); Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-1.67 to 2.20], Standard Error of Mean 0.99

3. Primary Outcome: 90-Day Hospital Readmission Rate
Description: 90-Day Readmissions will be measured using an all-cause readmission rate from inpatient claims for physical and behavioral health service use within 90 days following discharge from the qualifying inpatient admission prior to enrollment in the study.
Time Frame: 1 to 90 days
Population: 8 participants (0.57%) have missing readmission data. Since 31 participants had more than one admission within 90 days, a binary indicator of readmission within 90 days was generated and used as a primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 557 | 541 | 281
Participants
  No readmission within 90 days | 472 | 470 | 240
  At least one readmission within 90 days | 85 | 71 | 41
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall Test of Marginal Group Differences; Test type: Superiority; p = 0.59, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-squared statistics 0.08 with degrees of freedom (2)
Statistical Analysis 2: Comparison: High-Touch vs Optimal Discharge Planning; Test for the Treatment Effect; Test type: Superiority; p = 0.6692, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-square statistics 0.8 with degrees of freedom (2); Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.76 to 2.11]
Statistical Analysis 3: Comparison: High-Tech vs Optimal Discharge Planning; Test for the Treatment Effect; Test type: Superiority; p = 0.6692, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-square statistics 0.80 with degrees of freedom (2); Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.70 to 1.93]
Statistical Analysis 4: Comparison: High-Touch vs High-Tech; Test for the Treatment Effect; Test type: Superiority; p = 0.6692, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-square statistics 0.8 with degrees of freedom (2); Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.75 to 1.59]

4. Secondary Outcome: 30-Day Hospital Readmission Rate
Description: 30-Day Readmissions will be measured using an all-cause readmission rate in claims for physical and behavioral health service use within 30 days following discharge from the qualifying inpatient admission prior to enrollment in the study.
Time Frame: 1 to 30 days
Population: Since only 2 participants had more than one admission (2 admissions) within 30 days, a binary indicator of readmission within 30 days was generated and used as the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 559 | 545 | 283
Participants
  No readmission within 30 days | 535 | 528 | 272
  At least one readmission within 30 days | 24 | 17 | 11
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall Test of Marginal Group Differences; Test type: Superiority; p = 0.58, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-squared statistics 0.08 with degrees of freedom (2)
Statistical Analysis 2: Comparison: High-Touch vs Optimal Discharge Planning; Test for the treatment effect; Test type: Superiority; p = 0.7436, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-squared statistics 0.59 with degrees of freedom (2); Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.43 to 3.02]
Statistical Analysis 3: Comparison: High-Tech vs Optimal Discharge Planning; Test for the treatment effect; Test type: Superiority; p = 0.7436, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-squared statistics 0.59 with degrees of freedom (2); Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.31 to 2.25]
Statistical Analysis 4: Comparison: High-Touch vs High-Tech; Test for the treatment effect; Test type: Superiority; p = 0.7436, Regression, Logistic; Chi-squared statistics 0.59 with degrees of freedom (2); Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.62 to 2.97]

5. Secondary Outcome: Functional Status
Description: Assessed using the PROMIS Physical Function - Short Form 6b with six self-reported physical function measures to assess current function, including activities of daily living. Each question has five response options (a 5-point Likert scale) ranging from one to five with 5 being the highest level of physical function and 1 being the lowest. Per best practices, the instrument is scored by Health Measures Scoring Service, using item-level calibrations using responses to each item for each participant, producing a T-score. The highest possible T-score score is 59, indicating the highest level of physical function, and the lowest is 21, indicating the lowest level of physical function.
Time Frame: Baseline, 3-, 6-, and 12-months.
Population: Includes all individuals who completed the measure at least one timepoint.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 478 | 494 | 224
T score
  Baseline | 36.75 (7.89) | 36.29 (7.98) | 35.78 (7.60)
  3-Month: number analyzed (Participants) | 442 | 468 | 215
  3-Month | 37.11 (7.65) | 37.02 (7.97) | 36.83 (8.20)
  6-Month: number analyzed (Participants) | 422 | 445 | 205
  6-Month | 37.30 (7.87) | 36.85 (7.76) | 37.24 (7.91)
  12-Month: number analyzed (Participants) | 427 | 439 | 209
  12-Month | 36.99 (8.65) | 36.73 (8.14) | 36.29 (7.66)
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall test of treatment-by-time interaction; Test type: Superiority; p = 0.5558, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.82 with degrees of freedom (6, 3057)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change over time when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 6.74 with degrees of freedom (3, 3063)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change by treatment when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.7846, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.24 with degrees of freedom (2,1197)
Statistical Analysis 4: Comparison: High-Touch vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12 months using the linear contrasts; Test type: Superiority; p = 0.2444, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-Statistics 1.36 with degrees of freedom (1, 3057); Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.92 to 0.49], Standard Error of Mean 0.61
Statistical Analysis 5: Comparison: High-Tech vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12 months using the linear contrasts; Test type: Superiority; p = 0.6480, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.21 with degrees of freedom (1, 3057); Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.48 to 0.92], Standard Error of Mean 0.61
Statistical Analysis 6: Comparison: High-Touch vs High-Tech; Test for Group difference in the change from baseline to 12 months using the linear contrasts; Test type: Superiority; p = 0.3476, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.88 with degrees of freedom (1, 3057); Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.34 to 0.47], Standard Error of Mean 0.46

6. Secondary Outcome: Quality of Life
Description: Quality of Life will be assessed using the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF), which is a self-report measure consisting of 16 questions designed to enable investigators to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning during the past week. The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score, ranging from 14 to 70. The raw total score is calculated into a maximum possible score using the following formula: (raw total score - minimum score)/(maximum possible raw score - minimum score). The minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70. Thus, the formula for maximum score can also be written as: (raw score - 14)/56.
Time Frame: Baseline, 3-, 6-, and 12-months.
Population: Includes all individuals who completed the measure at least one timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 492 | 504 | 236
score on a scale
  Baseline | 0.50 (0.19) | 0.51 (0.19) | 0.51 (0.21)
  3-Month: number analyzed (Participants) | 455 | 477 | 227
  3-Month | 0.52 (0.19) | 0.52 (0.19) | 0.52 (0.20)
  6-Month: number analyzed (Participants) | 436 | 454 | 215
  6-Month | 0.52 (0.20) | 0.52 (0.20) | 0.52 (0.21)
  12-Month: number analyzed (Participants) | 441 | 449 | 218
  12-Month | 0.54 (0.20) | 0.52 (0.19) | 0.53 (0.19)
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall test of treatment-by-time; Test type: Superiority; p = 0.5199, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.86 with degrees of freedom (6, 3148)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change over time when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.0008, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 5.56 with degrees of freedom (3, 3154)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change by treatment when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.9897, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.01 with degrees of freedom (2,1229)
Statistical Analysis 4: Comparison: High-Touch vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12 months using the linear contrasts; Test type: Superiority; p = 0.8749, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.02 with degrees of freedom (1, 3148); Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.03 to 0.03], Standard Error of Mean 0.01
Statistical Analysis 5: Comparison: High-Tech vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12 months using the linear contrasts; Test type: Superiority; p = 0.2216, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.49 with degrees of freedom (1, 3148); Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.05 to 0.01], Standard Error of Mean 0.01
Statistical Analysis 6: Comparison: High-Touch vs High-Tech; Test for Group difference in the change from baseline to 12 months using the linear contrasts; Test type: Superiority; p = 0.0607, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 3.52 with degrees of freedom (1, 3148); Mean Difference (Final Values) = 0.02, 95% CI 2-sided [0.00 to 0.04], Standard Error of Mean 0.01

7. Secondary Outcome: Care Satisfaction
Description: Care satisfaction will be assessed using the Patient Assessment of Care for Chronic Conditions (PACIC) Survey. The PACIC Survey consists of 20-items that measures specific actions or qualities of care that patients report they have experienced in the care of their chronic conditions over the past 6 months. Each item is measured on a scale from 1-5 with 5 signifying higher patient satisfaction and 1 being the lowest. Scoring requires obtaining the mean of all 20 items.
Time Frame: Baseline, 3-, 6-, and 12-months.
Population: Includes all individuals who completed the measure at least one timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 492 | 502 | 236
score on a scale
  Baseline | 2.96 (0.98) | 2.86 (0.94) | 2.96 (1.00)
  3-Month: number analyzed (Participants) | 452 | 477 | 227
  3-Month | 3.02 (1.00) | 2.99 (0.99) | 2.97 (0.97)
  6-Month: number analyzed (Participants) | 436 | 454 | 215
  6-Month | 3.03 (0.98) | 2.97 (1.01) | 2.93 (1.00)
  12-Month: number analyzed (Participants) | 436 | 446 | 215
  12-Month | 3.05 (1.01) | 3.03 (1.01) | 3.00 (0.99)
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall test of treatment-by-time; Test type: Superiority; p = 0.1884, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.46 with degrees of freedom (6, 3138)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change over time when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.0090, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 3.87 with degrees of freedom (3, 3144)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change by treatment when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.2170, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.53 with degrees of freedom (2, 1227)
Statistical Analysis 4: Comparison: High-Touch vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12 months using the linear contrasts; Test type: Superiority; p = 0.1910, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.71 with degrees of freedom (1, 3138); Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.06 to 0.28], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: High-Tech vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12 months using the linear contrasts; Test type: Superiority; p = 0.0229, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 5.18 with degrees of freedom (1, 3138); Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.03 to 0.35], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: High-Touch vs High-Tech; Test for Group difference in the change from baseline to 12 months using the linear contrasts; Test type: Superiority; p = 0.2547, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.30 with degrees of freedom (1, 3138); Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.21 to 0.06], Standard Error of Mean 0.07

8. Secondary Outcome: Emergent Care Use
Description: Emergent care use will be measured using existing behavioral and physical health claims data to determine the frequency of emergency department visits within 12-months from enrollment.
Time Frame: Assessed at baseline, 6- and 12-Months.
Population: For each timepoint, participants who were eligible for Medicaid/Medicaid-Medicare with available claims data during at least 9 months (non-continuous) of the past 12 months.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 551 | 535 | 274
visits
  Baseline: number analyzed (Participants) | 515 | 509 | 254
  Baseline | 2.83 (3.25) | 2.40 (3.36) | 2.39 (3.73)
  6-Month | 1.33 (2.08) | 1.31 (2.44) | 1.25 (2.02)
  12-Month: number analyzed (Participants) | 529 | 520 | 260
  12-Month | 2.41 (3.58) | 2.40 (4.32) | 2.29 (3.29)
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall test for the treatment-by-time interaction; Test type: Superiority; p = 0.0413, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 2.49 with degrees of freedom (4, 3164)
Statistical Analysis 2: Comparison: High-Touch vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.1433, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 2.14 with degrees of freedom (1, 3164); Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.28 to 0.04], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: High-Tech vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.4272, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.63 with degrees of freedom (1, 3164); Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.10 to 0.23], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: High-Touch vs High-Tech; Test for Group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.0037, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 8.45 with degrees of freedom (1, 3164); Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.31 to -0.06], Standard Error of Mean 0.06

9. Secondary Outcome: Engagement in Primary Care
Description: Engagement in primary care will be measured using existing behavioral and physical health claims determining participant frequency of non-acute visits for participants in the 12 months following enrollment. Because clinical standards of care are 1 primary care (PCP) visit every 12 months, PCP visits are assessed as a Y/N variable at 12-Months.
Time Frame: Assessed at baseline, 6- and 12-Months.
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 559 | 545 | 283
Participants
  Baseline: At least one PCP visit | 451 | 468 | 224
  Baseline: No PCP visit | 64 | 41 | 30
  Baseline: Missing Data | 44 | 36 | 29
  6-Months: At least one PCP visit | 467 | 463 | 242
  6-Months: No PCP visit | 84 | 72 | 32
  6-Months: Missing Data | 8 | 10 | 9
  12-Months: At least one PCP visit | 467 | 476 | 238
  12-Months: No PCP visit | 62 | 44 | 22
  12-Months: Missing Data | 30 | 25 | 23
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall test for the treatment-by-time interaction; Test type: Superiority; p = 0.8231, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.38 with degrees of freedom (4, 3164)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change over time when the treatment-by-time interaction effect is not significant; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 330.05 with degrees of freedom (2, 1948)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change by treatment when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.6061, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.50 with degrees of freedom (2 , 1948)
Statistical Analysis 4: Comparison: High-Touch vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.7459, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.11 with degrees of freedom (1, 3164); Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.15 to 0.11], Standard Error of Mean 0.05
Statistical Analysis 5: Comparison: High-Tech vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.3169, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.00 with degrees of freedom (1, 3164); Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.18 to 0.08], Standard Error of Mean 0.05
Statistical Analysis 6: Comparison: High-Touch vs High-Tech; Test for Group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.4098, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.68 with degrees of freedom (1, 3164); Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.07 to 0.14], Standard Error of Mean 0.04

10. Secondary Outcome: Engagement in Specialty Care
Description: Engagement in specialty care will be measured using existing behavioral and physical health claims data determining participant frequency of specialty provider visits for participants in the 12 months following enrollment. Specialty care is inclusive of any care provided outside of primary care, physical therapy, or occupational therapy.
Time Frame: Assessed at baseline, 6- and 12-Months.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 551 | 535 | 274
visits
  Baseline: number analyzed (Participants) | 515 | 509 | 254
  Baseline | 7.29 (10.20) | 7.54 (8.89) | 7.20 (8.50)
  6-Month | 4.15 (5.34) | 4.51 (6.53) | 4.08 (5.16)
  12-Month: number analyzed (Participants) | 529 | 520 | 260
  12-Month | 7.80 (9.02) | 8.31 (10.39) | 7.84 (9.33)
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall test for the treatment-by-time interaction; Test type: Superiority; p = 0.4732, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.88 with degrees of freedom (4, 1945)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change over time when the treatment-by-time interaction effect is not significant; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 319.14 with degrees of freedom (2, 1948)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change by treatment when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.9628, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.04 with degrees of freedom (2, 1948)
Statistical Analysis 4: Comparison: High-Touch vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.8438, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.04 with degrees of freedom (1, 1945); Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.16 to 0.19], Standard Error of Mean 0.07
Statistical Analysis 5: Comparison: High-Tech vs Optimal Discharge Planning; Test for Group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.7425, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.11 with degrees of freedom (1, 1945); Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.19 to 0.15], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: High-Touch vs High-Tech; Test for Group difference in the change from baseline to 12-Months using the linear contrasts; Test type: Superiority; p = 0.5044, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.45 with degrees of freedom (1, 1945); Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.10 to 0.17], Standard Error of Mean 0.06

11. Secondary Outcome: Inpatient Readmissions Over 12-Months
Description: Readmissions over 12 months will be measured using an all-cause readmission rate from inpatient claims for physical and behavioral health service use within one year following discharge from the qualifying inpatient admission prior to enrollment in the study. Inpatient readmissions were lower than hypothesized for the population. As such, we assessed a Y/N variable for inpatient readmissions at 12-Months.
Time Frame: Assessed at baseline, 6- and 12-Months.
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 559 | 545 | 283
Participants
  Baseline: No inpatient admission | 342 | 344 | 170
  Baseline: One or more inpatient admissions | 173 | 165 | 84
  Baseline: Missing Data | 44 | 36 | 29
  6-Month: No inpatient admission | 412 | 400 | 201
  6-Month: One or more inpatient admissions | 139 | 135 | 73
  6-Month: Missing Data | 8 | 10 | 9
  12-Month: No inpatient admission | 337 | 332 | 170
  12-Month: One or more inpatient admissions | 192 | 188 | 90
  12-Month: Missing Data | 30 | 25 | 23
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall test for the treatment-by-time interaction; Test type: Superiority; p = 0.9804, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.11 with degrees of freedom (4, 3164)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change over time when the treatment-by-time interaction effect is not significant; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 21.80 with degrees of freedom (2, 3168)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change by treatment when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.9764, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.02 with degrees of freedom (2, 1211)
Statistical Analysis 4: Comparison: High-Touch vs Optimal Discharge Planning; Odds ratio of Treatment at 12-Months; Test type: Superiority; p = 0.9757, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; T-test statistics 0.03; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.63 to 1.60]
Statistical Analysis 5: Comparison: High-Tech vs Optimal Discharge Planning; Odds ratio of Treatment at 12-Months; Test type: Superiority; p = 0.7958, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; T-test statistics 0.26; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.67 to 1.68]
Statistical Analysis 6: Comparison: High-Touch vs High-Tech; Odds ratio of Treatment at 12-Months; Test type: Superiority; p = 0.7646, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; T-statistics -0.30; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.67 to 1.34]

12. Secondary Outcome: Mental Health Care Visits
Description: Assessed using existing behavioral health claims data determining frequency of mental health care visits for participants in the 12 months following enrollment. Because of the low frequency, we assess mental health care visits as a Y/N variable.
Time Frame: Assessed at baseline, 6- and 12-Months.
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 559 | 545 | 283
Participants
  Baseline: No mental health care visits | 479 | 476 | 237
  Baseline: At least one mental health care visit | 36 | 33 | 17
  Baseline: Missing Data | 44 | 36 | 29
  6-Months: No mental health care visits | 527 | 506 | 256
  6-Months: At least one mental health care visit | 24 | 29 | 18
  6-Months: Missing Data | 8 | 10 | 9
  12-Months: No mental health care visits | 492 | 484 | 238
  12-Months: At least one mental health care visit | 37 | 36 | 22
  12-Months: Missing Data | 30 | 25 | 23
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Overall test for the treatment-by-time interaction; Test type: Superiority; p = 0.9622, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.15 with degrees of freedom (4, 3164)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change over time when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.0377, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 3.28 with degrees of freedom (2, 3168)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the change by treatment when the treatment-by-time interaction effect is not significant; Test type: Superiority; p = 0.8300, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistic 0.19 with degrees of freedom (2, 1903)
Statistical Analysis 4: Comparison: High-Touch vs Optimal Discharge Planning; Odds ratio of Treatment at 12-Months; Test type: Superiority; p = 0.7507, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; T-statistics -0.32; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.38 to 2.00]
Statistical Analysis 5: Comparison: High-Tech vs Optimal Discharge Planning; Odds ratio of Treatment at 12-Months; Test type: Superiority; p = 0.8844, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; T-statistics -0.15; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.42 to 2.13]
Statistical Analysis 6: Comparison: High-Touch vs High-Tech; Odds ratio of Treatment at 12-Months; Test type: Superiority; p = 0.8227, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; T-statistics -0.22; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.49 to 1.77]

13. Secondary Outcome: Gaps in Care: Asthma
Description: Gaps in care will be assessed using Healthcare Effectiveness Data and Information Set (HEDIS) quality metrics. For asthma, we assess the percentage of members 21-64 years of age during the measurement year who were identified as having persistent asthma and were dispensed appropriate medications that they remained on during the treatment period. Two rates are reported:
  1. The percentage of members who remained on an asthma controller medication for at least 50% of their treatment period (MMA-1a).
  2. The percentage of members who remained on an asthma controller medication for at least 75% of their treatment period (MMA-1b).
Time Frame: Assessed at baseline, 6- and 12-Months
Population: Only a very small portion of our total sample size was eligible for Gaps in Care analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 8 | 13 | 6
Participants
  Baseline MMA-1a (50%): Did not close gap in care | 6 | 3 | 3
  Baseline MMA-1a (50%): Closed gap in care | 2 | 10 | 3
  6-Month MMA-1a (50%): number analyzed (Participants) | 4 | 11 | 3
  6-Month MMA-1a (50%): Did not close gap in care | 2 | 3 | 1
  6-Month MMA-1a (50%): Closed gap in care | 2 | 8 | 2
  12-Month MMA-1a (50%): number analyzed (Participants) | 6 | 7 | 2
  12-Month MMA-1a (50%): Did not close gap in care | 1 | 1 | 0
  12-Month MMA-1a (50%): Closed gap in care | 5 | 6 | 2
  Baseline MMA-1b (75%): Did not close gap in care | 6 | 9 | 3
  Baseline MMA-1b (75%): Closed gap in care | 2 | 4 | 3
  6-Month MMA-1b (75%): number analyzed (Participants) | 4 | 11 | 3
  6-Month MMA-1b (75%): Did not close gap in care | 2 | 4 | 1
  6-Month MMA-1b (75%): Closed gap in care | 2 | 7 | 2
  12-Month MMA-1b (75%): number analyzed (Participants) | 6 | 7 | 2
  12-Month MMA-1b (75%): Did not close gap in care | 1 | 4 | 0
  12-Month MMA-1b (75%): Closed gap in care | 5 | 3 | 2
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Frequency and test of the marginal association between event rate and treatment for eligible participants' data at 12 months for MMA-1a; Test type: Other; p = 1.00, Fisher Exact; Fisher's exact test for the null hypothesis of no association between each event and treatment group
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Frequency and test of the marginal association between event rate and treatment for eligible participants' data at 12 months for MMA-1b; Test type: Other; p = 0.242, Fisher Exact; Fisher's exact test for the null hypothesis of no association between each event and treatment group

14. Secondary Outcome: Gaps in Care: Chronic Obstructive Pulmonary Disease (COPD)
Description: Gaps in care will be assessed using Healthcare Effectiveness Data and Information Set (HEDIS) quality metrics. For COPD, we assess the percentage of COPD exacerbations for members 40 years of age and older who had an acute inpatient discharge or ED encounter and who were dispensed appropriate medications. Two rates reported:
  1. Dispensed a systemic corticosteroid within 14 days of the event (PCE-1)
  2. Dispensed a bronchodilator within 30 days of the event (PCE-2)
Time Frame: Assessed at baseline, 6- and 12-Months
Population: Only a very small portion of the total sample was eligible for COPD Gaps in Care analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 57 | 54 | 23
Participants
  Baseline PCE-1: number analyzed (Participants) | 24 | 28 | 15
  Baseline PCE-1: Did not close gap in care | 4 | 3 | 1
  Baseline PCE-1: Closed gap in care | 20 | 25 | 14
  6-Month PCE-1: Did not close gap in care | 8 | 2 | 1
  6-Month PCE-1: Closed gap in care | 49 | 52 | 22
  12-Month PCE-1: number analyzed (Participants) | 35 | 34 | 14
  12-Month PCE-1: Did not close gap in care | 2 | 1 | 3
  12-Month PCE-1: Closed gap in care | 33 | 33 | 11
  Baseline PCE-2: number analyzed (Participants) | 24 | 28 | 15
  Baseline PCE-2: Did not close gap in care | 8 | 4 | 3
  Baseline PCE-2: Closed gap in care | 16 | 24 | 12
  6-Month PCE-2: Did not close gap in care | 7 | 8 | 3
  6-Month PCE-2: Closed gap in care | 50 | 46 | 20
  12-Month PCE-2: number analyzed (Participants) | 35 | 34 | 14
  12-Month PCE-2: Did not close gap in care | 5 | 7 | 1
  12-Month PCE-2: Closed gap in care | 30 | 27 | 13
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test of the marginal association between event rate and treatment for eligible participants' data at 12 months for PCE-1; Test type: Other; p = 0.1112, Fisher Exact; Fisher's exact test for the null hypothesis of no association between each event and treatment group
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test of the marginal association between event rate and treatment for eligible participants' data at 12 months for PCE-2; Test type: Other; p = 0.4754, Fisher Exact; Fisher's exact test for the null hypothesis of no association between each event and treatment group

15. Secondary Outcome: Gaps in Care: Congestive Heart Failure (CHF)
Description: For Gaps in care related to CHF, we assess readmission rate within 30 days after discharge from inpatient stay for members with a diagnosis of CHF prior index hospitalization.
Time Frame: Assessed at 30-days from an index admission discharge.
Population: Only a small portion of the total sample was eligible for CHF Gaps in Care analyses.
Measure: Mean (Standard Deviation); unit: Number of readmissions within 30 days
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 84 | 98 | 39
Number of readmissions within 30 days
  Baseline: number analyzed (Participants) | 76 | 93 | 37
  Baseline | 0.04 (0.17) | 0.04 (0.17) | 0.02 (0.11)
  6-Month | 0.02 (0.10) | 0.04 (0.15) | 0.03 (0.12)
  12-Month: number analyzed (Participants) | 79 | 95 | 36
  12-Month | 0.04 (0.13) | 0.04 (0.13) | 0.04 (0.12)
Statistical Analysis 1: Comparison: High-Touch vs Optimal Discharge Planning; Test for the treatment effect (without weight) using a Firth's penalized logistic regression model for rare events; Test type: Superiority; p = 0.9079, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-squared statistics 0.19 with degrees of freedom (2); Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.13 to 4.28]
Statistical Analysis 2: Comparison: High-Tech vs Optimal Discharge Planning; Test for the treatment effect (without weight) using a Firth's penalized logistic regression model for rare events; Test type: Superiority; p = 0.9079, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-squared statistics 0.19 with degrees of freedom (2); Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.13 to 3.72]
Statistical Analysis 3: Comparison: High-Touch vs High-Tech; Test for the treatment effect (without weight) using a Firth's penalized logistic regression model for rare events; Test type: Superiority; p = 0.9079, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Chi-squared statistics 0.19 with degrees of freedom (2); Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.34 to 3.45]

16. Secondary Outcome: Gaps in Care: Cardiovascular Disease (CVD)
Description: Gaps in care will be assessed using Healthcare Effectiveness Data and Information Set (HEDIS) quality metrics. For CVD, we assess the percentage of males 21-75 years of age and females 40-75 years of age during the measurement year, who were identified as having clinical atherosclerotic cardiovascular disease (ASCVD) and met the following criteria. The following rates are reported:
  1. Received Statin Therapy. Members who were dispensed at least one high-intensity or moderate-intensity statin medication during the measurement year (SPC-1).
  2. Statin Adherence 80%. Members who remained on a high-intensity or moderate-intensity statin medication for at least 80% of the treatment period (SPC-2).
Time Frame: Assessed at baseline, 6- and 12-Months
Population: Only a very small portion of the total sample was eligible for CVD Gaps in Care analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 59 | 79 | 40
Participants
  Baseline SPC-1: number analyzed (Participants) | 45 | 42 | 27
  Baseline SPC-1: Did not close gap in care | 7 | 4 | 5
  Baseline SPC-1: Closed gap in care | 38 | 38 | 22
  6-Month SPC-1: number analyzed (Participants) | 50 | 54 | 32
  6-Month SPC-1: Did not close gap in care | 8 | 5 | 6
  6-Month SPC-1: Closed gap in care | 42 | 49 | 26
  12-Month SPC-1: Did not close gap in care | 11 | 10 | 7
  12-Month SPC-1: Closed gap in care | 48 | 69 | 33
  Baseline SPC-2: number analyzed (Participants) | 38 | 38 | 22
  Baseline SPC-2: Did not close gap in care | 16 | 6 | 7
  Baseline SPC-2: Closed gap in care | 22 | 32 | 15
  6-Month SPC-2: number analyzed (Participants) | 42 | 49 | 26
  6-Month SPC-2: Did not close gap in care | 11 | 17 | 11
  6-Month SPC-2: Closed gap in care | 31 | 32 | 15
  12-Month SPC-2: number analyzed (Participants) | 48 | 69 | 33
  12-Month SPC-2: Did not close gap in care | 14 | 23 | 14
  12-Month SPC-2: Closed gap in care | 34 | 46 | 19
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the treatment-by-time interaction (without weight) for SPC-1; Test type: Superiority; p = 0.9912, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.07 with degrees of freedom (4, 335)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change over time for SPC-1; Test type: Superiority; p = 0.8760, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.13 with degrees of freedom (2, 339)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change in treatment effect for SPC-1; Test type: Superiority; p = 0.6780, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.39 with degrees of freedom (2, 276)
Statistical Analysis 4: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the treatment-by-time interaction (without weight) for SPC-2; Test type: Superiority; p = 0.1761, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.59 with degrees of freedom (4, 284)
Statistical Analysis 5: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change over time for SPC-2; Test type: Superiority; p = 0.3239, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.13 with degrees of freedom (2, 288)
Statistical Analysis 6: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change in treatment effect for SPC-2; Test type: Superiority; p = 0.7415, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.30 with degrees of freedom (2, 139)

17. Secondary Outcome: Gaps in Care: Diabetes
Description: Gaps in care will be assessed using Healthcare Effectiveness Data and Information Set (HEDIS) quality metrics. For diabetes, we assess the percentage of members 40-75 years of age during the measurement year with diabetes who do not have clinical atherosclerotic cardiovascular disease (ASCVD) who met the following criteria. Two rates are reported:
  1. Received Statin Therapy. Members who were dispensed at least one statin medication of any intensity during the measurement year (SPD-1).
  2. Statin Adherence 80%. Members who remained on a statin medication of any intensity for at least 80% of the treatment period (SPD-2).
Time Frame: Assessed at baseline, 6- and 12-Months
Population: Only a very small portion of the total sample was eligible for Diabetes Gaps in Care analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 107 | 119 | 59
Participants
  Baseline SPD-1: number analyzed (Participants) | 105 | 119 | 59
  Baseline SPD-1: Did not close gap in care | 25 | 24 | 15
  Baseline SPD-1: Closed gap in care | 80 | 95 | 44
  6-Month SPD-1: number analyzed (Participants) | 107 | 104 | 45
  6-Month SPD-1: Did not close gap in care | 28 | 25 | 12
  6-Month SPD-1: Closed gap in care | 79 | 79 | 33
  12-Month SPD-1: number analyzed (Participants) | 88 | 88 | 34
  12-Month SPD-1: Did not close gap in care | 20 | 19 | 9
  12-Month SPD-1: Closed gap in care | 68 | 69 | 25
  Baseline SPD-2: number analyzed (Participants) | 80 | 95 | 44
  Baseline SPD-2: Did not close gap in care | 19 | 31 | 18
  Baseline SPD-2: Closed gap in care | 61 | 64 | 26
  6-Month SPD-2: number analyzed (Participants) | 79 | 79 | 33
  6-Month SPD-2: Did not close gap in care | 18 | 27 | 11
  6-Month SPD-2: Closed gap in care | 61 | 52 | 22
  12-Month SPD-2: number analyzed (Participants) | 68 | 69 | 25
  12-Month SPD-2: Did not close gap in care | 14 | 26 | 6
  12-Month SPD-2: Closed gap in care | 54 | 43 | 19
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the treatment-by-time interaction (without weight) for SPD-1; Test type: Superiority; p = 0.9786, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.11 with degrees of freedom (4, 608)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change over time for SPD-1; Test type: Superiority; p = 0.4703, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.76 with degrees of freedom (2, 612)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change in treatment effect for SPD-1; Test type: Superiority; p = 0.8770, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.13 with degrees of freedom (2, 332)
Statistical Analysis 4: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the treatment-by-time interaction (without weight) for SPD-2; Test type: Superiority; p = 0.6198, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.66 with degrees of freedom (4, 469)
Statistical Analysis 5: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change over time for SPD-2; Test type: Superiority; p = 0.6211, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.48 with degrees of freedom (2, 473)
Statistical Analysis 6: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change in treatment effect for SPD-2; Test type: Superiority; p = 0.1471, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.93 with degrees of freedom (2, 219)

18. Secondary Outcome: Gaps in Care: Depression
Description: Gaps in care will be assessed using Healthcare Effectiveness Data and Information Set (HEDIS) quality metrics. For depression, we assess the percentage of members diagnosed with a new episode of major depression, treated with antidepressant medication, and who remained on an antidepressant medication for:
  1. Effective Acute Phase Treatment - 84 days of continuous treatment during 114-day period following the Index Prescription Start Date (AMM-1).
  2. Effective Continuation Phase Treatment - 180 days of continuous treatment during 231-day period following the Index Prescription Start Date (AMM-2).
Time Frame: Assessed at baseline, 6- and 12-Months
Population: Only a very small portion of the total sample was eligible for Depression Gaps in Care analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
Number analyzed (Participants) | 56 | 59 | 34
Participants
  Baseline AMM-1: number analyzed (Participants) | 53 | 47 | 23
  Baseline AMM-1: Did not close gap in care | 24 | 12 | 10
  Baseline AMM-1: Closed gap in care | 29 | 35 | 13
  6-Month AMM-1: number analyzed (Participants) | 55 | 44 | 25
  6-Month AMM-1: Did not close gap in care | 20 | 14 | 6
  6-Month AMM-1: Closed gap in care | 35 | 30 | 19
  12-Month AMM-1: Did not close gap in care | 22 | 22 | 9
  12-Month AMM-1: Closed gap in care | 34 | 37 | 25
  Baseline AMM-2: number analyzed (Participants) | 53 | 47 | 23
  Baseline AMM-2: Did not close gap in care | 28 | 19 | 16
  Baseline AMM-2: Closed gap in care | 25 | 28 | 7
  6-Month AMM-2: number analyzed (Participants) | 55 | 44 | 25
  6-Month AMM-2: Did not close gap in care | 26 | 24 | 9
  6-Month AMM-2: Closed gap in care | 29 | 20 | 16
  12-Month AMM-2: Did not close gap in care | 32 | 31 | 14
  12-Month AMM-2: Closed gap in care | 24 | 28 | 20
Statistical Analysis 1: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the treatment-by-time interaction (without weight) for AMM-1; Test type: Superiority; p = 0.8247, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.38 with degrees of freedom (4, 280)
Statistical Analysis 2: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change over time for AMM-1; Test type: Superiority; p = 0.6651, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.41 with degrees of freedom (2, 284)
Statistical Analysis 3: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change in treatment effect for AMM-1; Test type: Superiority; p = 0.3441, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 1.07 with degrees of freedom (2, 218)
Statistical Analysis 4: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for the treatment-by-time interaction (without weight) for AMM-2; Test type: Superiority; p = 0.0847, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 2.07 with degrees of freedom (4, 280)
Statistical Analysis 5: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change over time for AMM-2; Test type: Superiority; p = 0.9695, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.03 with degrees of freedom (2, 284)
Statistical Analysis 6: Comparison: High-Touch vs High-Tech vs Optimal Discharge Planning; Test for change in treatment effect for AMM-2; Test type: Superiority; p = 0.9396, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F-statistics 0.06 with degrees of freedom (2, 200)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant 12 months following enrollment in the study.
Description: One High-Tech participant had 12-month claims outcomes and therefore was included in analysis although they were reported to the study team as being deceased (via self-report over the phone from a family member) and subsequently reported to the IRB as deceased at the final data collection timepoint. This participant is accounted for in under all-cause mortality and serious adverse events.
Arm/Group | High-Touch | High-Tech | Optimal Discharge Planning
All-Cause Mortality (participants affected / at risk) | 15/559 | 17/545 | 11/283
Serious Adverse Events (participants affected / at risk) | 0/559 | 0/545 | 0/283
Other Adverse Events (participants affected / at risk) | 0/559 | 0/545 | 0/283

LIMITATIONS AND CAVEATS:
Approximately 10% of our total sample was eligible for the gaps in care analysis using Healthcare Effectiveness Data and Information Set (HEDIS) data, and therefore, several HEDIS based outcomes were not adequately powered to demonstrate statistical significance.

Due to privacy and data sharing policies, we recognize not all claims related substance use diagnoses or behavioral health were obtained for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03451630/Prot_SAP_000.pdf